CLINICAL TRIAL: NCT06041373
Title: Verily Watch Cardio (AF and ECG) Study
Status: Withdrawn | Type: Observational
Why Stopped: It was decided by Verily Leadership to not pursue the study any further.
Sponsor: Verily Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 104343
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Paroxysmal Atrial Fibrillation Patients
  Interventions: Device: Verily Watch Cardio; Device: iRhythm Zio monitor; Device: Schiller CARDIOVIT FT-1

INTERVENTIONS:
Device: Verily Watch Cardio — The Verily Watch Cardio is an investigational wrist-worn wearable device containing multiple sensors to measure physiological and environmental metrics, including electrodes that enable a single-lead electrocardiogram (ECG) measurement and a photoplethysmogram (PPG) sensor to monitor for irregular pulses.
Device: iRhythm Zio monitor — The iRhythm Zio monitor, the reference device, is an FDA-cleared single-patient use, continuously recording ECG monitor that can be worn for up to 14 days.
Device: Schiller CARDIOVIT FT-1 — The Schiller CARDIOVIT FT-1, the reference device, is an FDA-cleared portable 12-lead ECG machine capable of recording continuous standard 12-lead resting ECG for up to 4 minutes.

SUMMARY:
This study is designed to evaluate the performance of the Verily Watch Cardio for recording electrocardiogram (ECG) and photoplethysmography (PPG) signals and detecting suspected atrial fibrillation (AF) episodes, in a free-living environment, in participants at risk for having an AF event.

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years old
* Able to read and speak English
* Participant understands the study requirements and is able and willing to sign written Informed Consent
* At risk of having an AF event, as determined by having a diagnosis of paroxysmal AF (PAF) and meeting one or more of the following:

  1. Scheduled or to be scheduled to undergo AF ablation
  2. AF burden of ≥25% in the 3 months prior to consent date as confirmed via an implantable loop recorder (ILR), holter monitor, or adhesive monitoring patch
  3. CHA2DS2VASc score ≥3
  4. Left atrial diameter ≥4.4 cm as confirmed by transthoracic echo (TTE) within one year of consent
* Without significant limitation in ability to participate in the study, in the opinion of the Investigator

Exclusion Criteria:

* Have a pacemaker or implantable cardioverter defibrillator (ICD)
* Currently on class Ic or class III antiarrhythmic medication that has been successful in eliminating AF (no documented AF of more than 30 seconds since the initiation of the medication). Should be at least one week off medication.
* Had successful AF ablation (no documented AF of more than 30 seconds post procedure)
* Known severe allergy to nickel or metal jewelry
* Known allergic reaction to polyester, nylon, spandex, adhesives or hydrogels; or with family history of adhesive skin allergies
* Are diagnosed with persistent AF
* Have an implantable neuro-stimulator
* Currently wearing an ECG patch that prevents the use of the FDA-cleared wearable ECG patch, at the discretion of the Investigator.
* Have discolored wrists (e.g., tattoos, ink), at the discretion of the Investigator.

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: At risk of having an AF event determined by a diagnosis of paroxysmal atrial fibrillation (PAF)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of suspected AF episode detection | Up to 14 days
  Sensitivity and Specificity of suspected AF episode detection by the irregular pulse detection algorithm

SECONDARY OUTCOMES:
A sensitivity analysis estimating the range of sensitivities and specificities | Up to 14 days
  A sensitivity analysis estimating the range of sensitivities and specificities observed when imputing missing test device data
Sensitivity and Specificity in defined subgroups | Up to 14 days
  Sensitivity and Specificity in subgroups defined by: race, age-groups, activity level, skin-tone and AF-burden
Mean difference in Interbeat interval (IBI) and the associated limits of agreement (LoA) | Up to 14 days
  Mean difference in Interbeat interval (IBI) and the associated limits of agreement (LoA) based on recorded ECG data
Participant-level and heartbeat level sensitivity/specificity of P-wave detection | Up to 14 days
  Participant-level and heartbeat level sensitivity/specificity of P-wave detection based on recorded ECG data

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ghanbari, MD, Principal Investigator — Verily Life Sciences
Locations (3):
- United States (3):
  - Colorado Heart and Vascular, Lakewood, Colorado
  - Ascension Providence Hospital, Southfield, Michigan
  - Wake Forest Medical Center, Winston-Salem, North Carolina